CLINICAL TRIAL: NCT04378751
Title: Promoting Genetic Counseling Among African American Women With a Family History of Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Vida Henderson, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2020-0342; K01CA248852-01 (NIH)
Record Dates: First submitted 2020-05-01; First posted 2020-05-07 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: High Risk for Breast Cancer

STUDY DESIGN:
Intervention Model Description: Computer-generated randomization (equal numbers in each arm), patients will be randomized to one of two arms:
  1. Decision aid video
  2. Genetic counseling informational brochure
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision aid video (Experimental): Participants receiving the intervention will complete a pretest, watch the decision aid video, and complete posttest via tablet computer facilitated by Patient Navigators.
  Interventions: Behavioral: Decision aid video
- Genetic counseling informational brochure (Active Comparator): Participants receiving the control will complete pretest, review a genetic counseling brochure with the Patient Navigators, and complete posttest via tablet computer facilitated by a Patient Navigator.
  Interventions: Behavioral: Genetic counseling informational brochure

INTERVENTIONS:
Behavioral: Decision aid video — Decision aid video
  Arms: Decision aid video
Behavioral: Genetic counseling informational brochure — Genetic counseling informational brochure
  Arms: Genetic counseling informational brochure

SUMMARY:
In the United States, carriers of hereditary genetic mutations have up to an 85% risk of developing breast cancer compared to 12% in the general population. Overall uptake of genetic services is generally low, particularly among high-risk African American (AA) women, who carry a disproportionate burden of breast cancer mortality. Further, although testing close relatives of individuals who test positive for a pathogenic variant might curtail breast cancer disparities attributable to hereditary risk, it is unclear how counseled or tested individuals influence their social and familial networks. Using a randomized control trial design, the objective of this research project is to test the effectiveness of a culturally targeted video, previously developed by our research team, on promoting genetic counseling attendance among AA women determined to be at high risk for breast cancer through cancer genetic risk assessment in a clinical setting. This study will also test how psychosocial factors (knowledge, intrinsic motivation, risk perception, and distress) impact the relationships between intervention exposures (video versus brochure) and compare the impact of intervention exposures on diffusion of knowledge about genetic counseling through social network analysis.

DETAILED DESCRIPTION:
Study Design. The investigator will conduct a randomized control trial single-blind control trial to test the effectiveness of a culturally targeted decision aid video to promote genetic counseling among African American determined to be high risk for breast cancer through cancer genetic risk assessment. Eligible patients will be randomly assigned to receive information about genetic counseling using a culturally targeted decision aid video (treatment group) or a brochure (control).

Research Protocol. As part of standard of care, patients will complete a cancer genetic risk assessment (CGRA) as part of intake on a tablet computer provided by the front desk clinic staff. CGRA results will be uploaded to the EMR, printed and given to a patient navigator. The patient navigator will approach patients, give them a recruitment flyer, information about the study, screen patients and obtain informed consent for women who choose to participate in the study. Based on computer-generated randomization (equal numbers in each arm), patients will be randomized to one of two groups to receive: 1) pretest, view decision aid video, and posttest or 2) pretest, genetic counseling brochure, and posttest. Both arms will be facilitated by patient navigators. Upon completion of posttest, patient navigators will ask women if they would like to make an appointment for genetic counseling, contact the provider for the order if not already in the EMR, make genetic counseling appointments for women who choose to attend, and monitor and collect follow-up data. All enrolled participants will receive a phone call at 4 weeks post-intervention to (a) verify counseling attendance through self-report and EMR extraction if applicable; (b) ask whether the patient was referred to genetic testing after her genetic counseling if applicable; and (c) ask whether other family members were referred to genetic services if applicable and (d) determine who in their social networks, if anyone, the participant told about genetic counseling, and if so, how this information was shared.

ELIGIBILITY:
Inclusion Criteria:

1. Are female
2. Identify as African American
3. Are age 25 or older
4. Speak and understand English
5. Completed a cancer genetic risk assessment (CGRA) as part of clinic intake
6. Are classified as high risk for developing breast cancer per CGRA
7. Have not previously received genetic counseling

Exclusion Criteria:

1. Are not female
2. Do not identify as African American
3. Are age 24 or younger
4. Do not speak and understand English
5. Did not complete a cancer genetic risk assessment (CGRA) as part of clinic intake
6. Are not classified as high risk for developing breast cancer per CGRA
7. Have previously received genetic counseling

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 80 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Genetic Counseling Attendance | 52 weeks
  Compare the effects of intervention vs. control arm on genetic counseling attendance among African American women recommended for genetic counseling through cancer genetic risk assessment.
  Assessed via EMR and survey at follow-up.
  2-item (Did patient complete genetic counseling appointment? A) Self-report and B) EMR)
  1 items assessing familial referral to genetic counseling or testing

SECONDARY OUTCOMES:
Decision Aid Usability | 52 weeks
  5-item agreement likert scale to assess usability, satisfaction, decisional conflict (e.g., I felt I could relate to what the actors were saying?)
  Assessed via survey at immediate posttest
Knowledge about Genetic Counseling | 52 weeks
  Items to assess changes in knowledge about genetic counseling for breast cancer risk between pre and post intervention; (e.g., A purpose of genetic counseling is to help people understand their options for genetic testing.)
  Relevant items from published instrument (Maio) and Facing Our Risk of Cancer Empowerment (FORCE) brochure (control arm brochure) adapted for genetic counseling for breast cancer.
  Assessed via survey at pretest and posttest.
Distress Associated with Genetic Counseling and Breast Cancer Risk | 52 weeks
  Items to assess patient worry/anxiety related to genetic counseling and breast cancer risk; (e.g., How often have you thought about your chances of getting cancer?)
  7-item Cancer Worry Scale
  Assessed via survey at pretest and posttest.
Intrinsic Motivation for Genetic Counseling Attendance | 52 weeks
  Items to assess motivation for genetic counseling attendance (e.g., The reason I would attend genetic counseling is because I feel that I want to take responsibility for my own health.)
  15-item Treatment Self-Regulation Questionnaire and 4-item Self-Efficacy Scale
  Assessed via survey at pretest and posttest.
Risk Perception Associated with Breast Cancer | 52 weeks
  Items to assess perception of risk related to getting breast cancer (In your opinion, compared to other women your age, what are your chances of getting breast cancer?)
  1-item question obtained from published instrument.
  Assessed via survey at pretest and posttest.
Diffusion of Knowledge | 56 weeks
  Items to assess sharing of knowledge among social and familial networks about genetic counseling. Diffusion of knowledge will be assessed by collecting data on social network size, composition, density, and information sharing related to genetic counseling and risks.
  Relevant social network assessment items-General Social Survey.
  Examples:
  * Name generator: (From time to time, most people discuss important matters with other people. Looking back over the past month, who are the people with whom you discussed genetic counseling or genetic risks?
  * Name interpreter: (e.g., What is relationship between you and X?)
  Assessed at 4 week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Kent Hoskins, MD, Principal Investigator — University of Illinois at Chicago
Locations (2):
- United States (2):
  - UIC Cancer Center, Chicago, Illinois
  - University of Illinois at Chicago Hospital and Ambulatory Clinics, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Undecided